CLINICAL TRIAL: NCT01187459
Title: Vitamin D in Pediatric Crohn's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H10-01391
Record Dates: First submitted 2010-08-20; First posted 2010-08-24 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Crohn's Disease; Dose Response
MeSH Terms: conditions — Vitamin D Deficiency; Crohn Disease | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10 ug/day (Experimental)
  Interventions: Dietary Supplement: Vitamin D
- 50 ug/day (Experimental)
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — 10 ug/day Vitamin D, taken for 6 months.
  Arms: 10 ug/day
Dietary Supplement: Vitamin D — 50 ug/day Vitamin D, taken for 6 months.
  Arms: 50 ug/day

SUMMARY:
Background: Crohn's disease (CD), a type of Inflammatory Bowel Disease (IBD), is a chronic relapsing inflammatory disorder of the digestive system. CD affects ~112,000 individuals in Canada, of whom 20-25% are diagnosed in childhood or adolescence. The specific cause of CD remains unknown; however, it is hypothesized that CD involves a complex interaction of several factors, including a genetically susceptible host, the intestinal mucosal immune system and microbe population. Several dietary factors have been explored for their potential role in the etiology of CD. However, no consensus on the role of diet has emerged. Recent evidence suggests a plausible link between a lack of Vitamin D and CD.

Purpose & Hypothesis: The investigators primary hypothesis is that a greater proportion of pediatric CD patients will achieve optimal 25OHD concentration (> 75 nmol/L) on 2000 IU/d than 400 IU/d Vitamin D.

Methods: Pediatric Crohn's Disease patients between 8-18 years of age, and have been in remission for at least 4 weeks as indicated by a Pediatric Crohn's Disease Activity Index (PCDAI) <10 will be recruited for a double-blind, randomized, controlled trial where they will receive one of two dosages of vitamin D (10 or 50 ug/day) and will be asked to continue the supplementation for 6 months. Vitamin D levels will be measured in blood at baseline, 3 months, and 6 months. Dietary vitamin D intake will be estimated using a food frequency and lifestyle questionnaire. Data will be analyzed using multiple regression analysis controlling for baseline values.

Expected Results and Conclusions: It is expected that a greater proportion of children receiving the 50 ug/day vitamin D supplement will achieve a blood vitamin level >75 nmol/L compared to children receiving 10 ug/day. This data will aid policy makers, parents/children and healthcare workers in recommending an appropriate vitamin D dosage for the pediatric crohn's population.

DETAILED DESCRIPTION:
Trial Objectives: Our primary hypothesis is that a greater proportion of pediatric CD patients will achieve optimal 25OHD concentration (> 75 nmol/L) on 2000 IU/d than 400 IU/d Vitamin D. Our primary objective is to determine whether the proportion of pediatric CD patients achieving 25OHD concentration > 75 nmol/L is greater in those receiving 2000 IU/d or 400 IU/d Vitamin D. Our secondary objective is to determine if patients receiving 2000 IU Vitamin D are more likely to have remained in remission [Pediatric Crohn's Disease Activity Index (PCDAI) < 20] than those receiving 400 IU/d.

Study Design: This will be a parallel study design with two levels of Vitamin D: 400 IU/d, and 2000 IU/d supplement of Vitamin D3.

Study Duration: 6 Months

Number of Sites (inside and outside of Canada):

1. Children's and Women's Hospital of British Columbia
2. McMaster's Children's Hospital

List of Investigators:

* Tim Green, PhD. Faculty of Land and Food Systems, UBC
* Kevan Jacobson MD. Pediatric GI, UBC
* Robert Issenman MD. Pediatric GI, McMaster University
* Susan Barr PhD. Faculty of Land and Food Systems, UBC Sample Size: Forty-five subjects per group will allow us to detect as little as a 20% difference in the proportion of participants achieving a 25OHD >75 nmol/L between the two doses with 80% power and a one sided of 0.05. Assuming a 10% attrition rate we will need to recruit 50 subjects per group. Clinical experience indicates that approximately 50% of pediatric CD patients will relapse over 6 months based on an elevated PCDAI (>20). Forty-five subjects per group will allow us to detect a 50% difference in CD relapse between the two doses with 80% power and a one sided of 0.05.

Patient Population: Pediatric CD patients who are patients of the pediatric gastroenterology services of BC and McMaster Children's Hospitals.

Inclusion Criteria: Patients will be eligible to participate if they have a diagnosis of CD, are between 8-18 years of age, and have been in remission for at least 4 weeks as indicated by a PCDAI <10.

Exclusion Criteria: Patients will be ineligible if they have active disease with a PCDAI > 10, taking corticosteroids, or taking more than 400 IU Vitamin D at enrollment.

NHP Formulation: Vitamin D at doses of 10 and 50 ug (400, and 2000 IU) 400 IU DIN #02231624 2000 IU Dosage Regimen: Patients will be randomly assigned to one of two supplemental doses of vitamin D3 (10, and 50 ug/d) Prestudy Screening and Baseline Evaluation: Patients and their parent/guardian who meet the inclusion criteria and who consent will be enrolled and assigned without bias to a dose group. A one-hour fasting blood sample and a spot urine collection will be collected, a PCDAI will be administered, and patients will complete a food frequency questionnaire (FFQ) that will include information on Vitamin D and calcium supplement use (including dose and duration) as well as a lifestyle and demographic questionnaire.

Treatment Visit: One-hour fasting blood and spot urine will be collected and the PCDAI will be administered at baseline, 3 months (+/- 1 week), and 6 months (+/- 1 week) after baseline. 25OHD concentrations are thought to stabilize after 8 weeks of supplementation at a constant dose.

Premature Withdrawal/Discontinuation Criteria: Discontinuation criteria for individual subjects include violation of any of the exclusion criteria, severe non-compliance with the protocol, or occurrence of adverse events that are judged to be severe enough for discontinuation. Subjects are also free to voluntarily discontinue the study at any time.

Rescue Medication: Regular dosage of 400 IU vitamin D Washout Period: None Dietary Assessment: Calcium and Vitamin D intake from food over the previous month will be estimated using a food frequency questionnaire validated for use in a variety of ethnic groups (From S Whiting; U Sask).

Pediatric Crohn's Disease Activity Index: The PCDAI will be used to assess the severity of disease. It consists of a patient recall, laboratory values, and a clinical examination. Scores below 10 indicate remission and scores above 20 indicate active disease (attached).

Laboratory Assessment: Erythrocyte Sedimentation Rate, serum calcium, serum albumin, serum creatinine, urinary calcium and urinary creatinine will be measured by the hospital pathology labs using standard procedures. Serum 25OHD, PTH will be measured using automated chemiluminescent assay system (Liaison, Diasorin) by BC Biolabs.

Efficacy Analysis: The proportion of patients achieving a 25OHD of 75 nmol/L on each of the dosages at 6 months will be compared using a Chi-squared test. Likewise the proportion of participants remaining in remission (PCDAI <20) will also be compared using a Chi-squared test. Data will initially be analyzed as intent-to-treat for all outcomes. In the case of dropouts or missing data the last observation will be carried-forward. A second analysis will be carried out for each outcome only using subjects with complete data and who were over 80% compliant in supplement use (as-treated analysis). Differences in the characteristics of the participants in the groups at baseline will be determined using Student's t-test for continuous and the chi-square test or Fisher's Exact Test for categorical variables.

Safety Analysis: Adverse events will be recorded according to Good Clinical Practice Guidelines and the guidelines of our university's human research ethics board. Adverse event occurrences will be compared descriptively between the treatment and placebo groups. Safety will also be assessed as part of the blood collection (Serum Ca and Serum PTH and Serum P).

Statistical Analysis: Data will initially be analyzed as intent-to-treat for all outcomes. In the case of dropouts or missing data the last observation will be carried-forward. A second analysis will be carried out for each outcome only using subjects with complete data and who were over 80% complaint in supplement use (as-treated analysis). Differences in the characteristics of the participants in the groups at baseline will be determined using Student's t-test for continuous and the chi-square test of Fisher's Exact Test for categorical variables. The primary endpoints will be the dosages at 3 months will be evaluated using a Chi-squared test. Dose response (as ug Vitamin D3 per nmol/L increase in 25OHD) in children will be determined using multiple regression analysis with 25OHD as the dependent variable, vitamin D dose entered as a continuous variable, and baseline vitamin D as a covariate.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible to participate if they have a diagnosis of CD, are between 8-18 years of age, and have been in remission for at least 4 weeks as indicated by a PCDAI <10.

Exclusion Criteria:

* Patients will be ineligible if they have active disease with a PCDAI > 10, taking corticosteroids, or taking more than 400 IU Vitamin D at enrollment.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 87 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The proportion of pediatric CD patients achieving optimal 25OHD concentration | 6 months
  To determine whether the proportion of pediatric CD patients achieving 25OHD concentration > 75 nmol/L different between groups.

SECONDARY OUTCOMES:
If patients receiving 2000 IU Vitamin D are more likely to have remained in remission | 6 months
  To determine if patients receiving 2000 IU Vitamin D are more likely to have remained in remission [Pediatric Crohn's Disease Activity Index (PCDAI) < 20] than those receiving 400 IU/d.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - BC Children's Hospital, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario

REFERENCES:
- [Derived] Wingate KE, Jacobson K, Issenman R, Carroll M, Barker C, Israel D, Brill H, Weiler H, Barr SI, Li W, Lyon MR, Green TJ. 25-Hydroxyvitamin D concentrations in children with Crohn's disease supplemented with either 2000 or 400 IU daily for 6 months: a randomized controlled study. J Pediatr. 2014 Apr;164(4):860-5. doi: 10.1016/j.jpeds.2013.11.071. Epub 2014 Jan 11. PMID 24423431